CLINICAL TRIAL: NCT05428891
Title: Image-guided Pleural Needle Biopsy or Medical Thoracoscopy: Which Method for Which Patient? A Randomized Controlled Trial
Brief Title: Image-guided Pleural Biopsy or Medical Thoracosocopy in Diagnosis of Pleural Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Muzaffer Metintas, Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 80558721/162
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Diagnosis of Pleural Diseases
Keywords: Pleura; Thoracoscopy; Pleural needle biopsy; Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Randomized prospective
Who Masked: Participant
Masking Description: Participants do not know which method will apply.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Only pleural effusion (Other): The patients with only pleural effusion on their CT scans.
  Interventions: Procedure: Abrams' needle pleural biopsy (IG-ANPB) versus medical thoracoscopy in the diagnosis of pleural diseases.
- Pleural effusion associated with pleural thickening or any other lesion like mass or nodules. (Other): The patients with pleural effusion associated with pleural thickening or any other lesion-like mass or nodules on their CT scans.
  Interventions: Procedure: Abrams' needle pleural biopsy (IG-ANPB) versus medical thoracoscopy in the diagnosis of pleural diseases.

INTERVENTIONS:
Procedure: Abrams' needle pleural biopsy (IG-ANPB) versus medical thoracoscopy in the diagnosis of pleural diseases. — We compare the diagnostic efficacy and safety of imaging-guided Abrams needle biopsy with medical thoracoscopy.
  Other Names: A diagnostic algorithm for pleural diseases.

SUMMARY:
Pleural diseases can occur due to numerous pathological conditions. The increasing prevalence of etiologic causes and aging population worldwide will make pleural diseases a growing problem in the coming years. As a result of this increase, the need for diagnostic investigations is also increasing. In recent years, the use of image-guided needle biopsies under ultrasound (US) or computed tomography (CT) and the increasing use of medical thoracoscopy (MT) have significantly increased the accuracy of diagnosis of pleural disease. There is not yet a generally accepted algorithm for invasive diagnosis of pleural disease, widely used in clinics, that determines which method should be used in which patient. It would be necessary and valuable to develop an algorithm based on imaging findings in particular to improve the diagnostic accuracy, safety, and cost of the procedure. The investigators aimed to test the algorithm in an interventional study to increase the level of evidence in this study.

DETAILED DESCRIPTION:
No consensus exists regarding which biopsy methods are appropriate for specific procedures. In this randomized prospective study, the investigators aimed to compare image guided - pleural biopsy using an Abrams' needle (IG-ANPB) with medical thoracoscopy (MT) according to the CT findings of the patients concerning both diagnostic yield and safety.

Between May 2017 and March 2022, 228 patients with exudative pleural effusion who the cytological analysis could not diagnose were included. All patients were separated into two groups regarding the CT findings: Only pleural effusion or pleural effusion with pleural thickening/lesion. In each group, the patients were randomized to either underwent IG-ANPB or underwent MT. The two groups were compared in terms of diagnostic sensitivity, accuracy, and complications.

ELIGIBILITY:
Inclusion Criteria:

Pleural effusion Malignant pleural diseases Pleurisy tuberculosis Benign pleural diseases

Exclusion Criteria:

Age less than 18 years, Parapneumonic effusion, Presence of other systemic diseases that could interfere radiological evaluation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of pleural biopsy methods for the diagnosis of pleural diseases. | 60 months
  To compare the diagnostic efficacy and safety of imaging-guided Abrams needle biopsy with medical thoracoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Metintas, Prof., Principal Investigator — Eskisehir Osmangazi University Medical Faculty Department of Chest Diseases
Locations (1):
- Eskisehir Osmangazi University Medical Faculty Department of Chest Diseases, Eskişehir, Tepebaşı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metintas M, Ak G, Yildirim H, Dundar E, Aydin N, Erginel S, Alatas F, Yilmaz S, Metintas S. Image-Assisted Pleural Needle Biopsy or Medical Thoracoscopy: Which Method for Which Patient? A Randomized Controlled Trial. Chest. 2024 Aug;166(2):405-412. doi: 10.1016/j.chest.2024.03.038. Epub 2024 Mar 28. PMID 38554817